CLINICAL TRIAL: NCT05934708
Title: Examining the Role of Female Endogenous Sex Hormones in Eccentric Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-23-00363
Record Dates: First submitted 2023-06-20; First posted 2023-07-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Response
Keywords: menstrual cycle; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low estrogen; low progesterone (Experimental): Participants will come in while on their period. During this time estrogen and progesterone concentrations are low.
  Interventions: Behavioral: Eccentric leg extension
- High estrogen; low progesterone (Experimental): Participants will come in just before ovulation, when estrogen concentrations are high and progesterone concentrations remain low.
  Interventions: Behavioral: Eccentric leg extension
- Medium estrogen; high progesterone (Experimental): Participants will come in just after ovulation when estrogen concentrations are at a medium level, and progesterone concentrations are high.
  Interventions: Behavioral: Eccentric leg extension

INTERVENTIONS:
Behavioral: Eccentric leg extension — Participants will complete a 10 x 10 eccentric leg extension on a Cybex Norm dynamometer. Upon arrival, participants will be asked their perceived readiness to perform on a 11 point numeric rating scale. Before the running protocol a baseline blood sample will be collected, as well as passive and active delayed onset muscle soreness (DOMS), a countermovement jump. Half way through each set (i.e., after the 5th repetition) participants will be asked to rank their level of difficulty on a 11 point OMNI Res scale. This will occur during each set. Participants will have follow up blood draws, measures of muscle function (i.e, jump height) and soreness measured immediately after and 24 and 48 hours post-exercise.

SUMMARY:
The fluctuating concentrations of female sex hormones, namely estrogen and progesterone may have an effect on the ability of the tissue to withstand challenging exercise conditions, such as eccentric exercise. These sex hormones have also been purported to influence the perceived difficulty of exercise. This study aims to uncover how the different estrogen and progesterone concentrations present throughout the menstrual cycle effect perceived readiness to perform, perceptions of difficulty, and different recovery metrics.

DETAILED DESCRIPTION:
Although nearly half of the population is female, less than 10% of research resources are allocated to understanding how their dynamic physiology impacts athletic readiness, performance, and recovery. The fluctuating concentrations of female sex hormones, namely estrogen and progesterone may have an effect on the ability of the tissue to withstand challenging exercise conditions, such as eccentric exercise. This study aims to uncover how the different estrogen and progesterone concentrations present throughout the menstrual cycle effect perceived readiness to perform, perceptions of difficulty, and the inflammatory environment and quantification of muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* BMI of 18.5-29.9 as a BMI below or above these cut points results in highly varied menstrual cycle lengths [15]
* Not taking contraception or other types of medication that could influence reproductive status
* Regular menstruation
* Non-pregnant
* Medically free from chronic diseases
* Novel to downhill running
* Weight greater than or equal to 110 lbs
* Not taking exogenous hormones
* Not suffering from known gynecological disease (i.e., PCOS, endometriosis, etc.) that may influence menstrual cycle regularity

Exclusion Criteria:

* Amenorrhea or oligomenorrhea
* Perimenopausal or menopausal
* Recreational or professional trail or downhill runner
* On a form of contraception
* Cardiac disability
* Pacemaker
* Arterial disease
* Uncontrolled hemorrhage
* Blood clots
* Pregnant or trying to become pregnant
* Cancerous lesions
* Sensory or mental impairment
* Unstable fractures
* Weight less than 110 lbs
* Suffering from gynecological disease (i.e., PCOS, endometriosis, etc.) that may influence menstrual cycle regularity
* Taking exogenous hormones

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants will be cis-gendered female. This is to control for the potential influence that differing hormonal profiles have on transgender and nonbinary female athletes.
Enrollment: 30 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Preparedness to perform | Pre exercise
  Perceived readiness will be measured on an 11 point numeric rating scale (NRS) with 0 being not ready at all, and 10 being most prepared
Rating of difficulty | 30 minutes
  Perceived difficulty will be measured on a 11 point numeric rating scale called the OMNI res throughout the duration of exercise.
Inflammatory markers | Change over time (pre/post, 24 hour, 48 hour)
  Inflammatory markers (IL-6, IL-8, TNF-alpha, and IL-10) will be measured in blood serum to understand how the concentration of estrogen changes the inflammatory response to damaging exercise.
Counter movement jump height | Change over time (pre/post, 24 hour, 48 hour)
  A countermovement jump (CMJ) will be performed on VALD ForceDecks to determine muscle function overtime.
Passive Delayed Onset Muscle Soreness (DOMS) | Change over time (pre/post, 24 hour, 48 hour)
  DOMS will be assessed as participants are stationary to assess their perception of muscle damage over time.
Active Delayed Onset Muscle Soreness (DOMS) | Change over time (pre/post, 24 hour, 48 hour)
  DOMS will be assessed as participants complete a wall sit to assess their perception of muscle soreness over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Exercise Research Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No